CLINICAL TRIAL: NCT07004595
Title: Evaluation of Frailty in Patients With Fibrosing Interstitial Lung Diseases: Prognostic and Therapeutic Impact
Acronym: FRAPID
Status: Not yet recruiting | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: AP_CM_001
Record Dates: First submitted 2025-01-17; First posted 2025-06-04 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Sarcopenia
Keywords: Fibrosing interstitial lung diseases;; frailty; sarcopenia
MeSH Terms: conditions — Sarcopenia; Frailty

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Evaluation of patient frailty — Quality of Life questionnaire

SUMMARY:
Fibrosing interstitial lung diseases (ILDs), with idiopathic pulmonary fibrosis being the most common form, primarily affect older individuals and have a poor prognosis, with a median survival of 3 to 5 years. While antifibrotic treatments such as nintedanib and pirfenidone can slow disease progression, their efficacy is often limited by side effects, particularly in elderly patients. A comprehensive patient assessment, including evaluations of frailty and sarcopenia, could optimize care by identifying those at risk for poor outcomes or poor treatment tolerance. Frailty, characterized by reduced physiological reserves, and sarcopenia, defined as a loss of muscle mass and strength, are both associated with increased mortality and morbidity risks. Although their individual impacts on fibrosing ILDs have been documented, the combined effect of these two syndromes on patient prognosis remains unexplored, highlighting the need for further studies to guide therapeutic decision-making.

DETAILED DESCRIPTION:
Frailty and sarcopenia are two distinct entities, each capable of worsening patient mortality and morbidity. Their association has been studied in the general population in a cohort of over 2,000 individuals aged 70 to 85 years (34816568). The prevalence of sarcopenia among frail participants was 40%. The characteristics and risks faced by patients who were both frail and sarcopenic differed from those who were only sarcopenic or only frail.

No study has evaluated the prognostic impact of the combined presence of sarcopenia and frailty on the outcomes of patients with fibrosing ILDs.

ELIGIBILITY:
Inclusion Criteria:

* Patient with fibrosing ILD according to the ATS/ERS/JRS/ALAT 2022 criteria.
* Patient aged ≥ 65 years.
* Outpatient consultation (scheduled appointment in an outpatient clinic, day hospital, or weekly hospital stay).
* French-speaking patient.
* Patient who has received an information sheet explaining the study and has not expressed opposition to participating in this research.

Exclusion Criteria:

* Patient under legal guardianship, curatorship, or judicial protection.
* Cognitive disorders limiting the use of questionnaires.
* Patient with a CT scan showing an early usual interstitial pneumonia (UIP) pattern according to the ATS/ERS/JRS/ALAT 2022 classification.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: The study population will consist of older adults who are incident cases of patients referred to Nantes University Hospital for the evaluation of fibrosing ILD
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-07-20 (Estimated); Primary Completion 2026-02-20 (Estimated); Study Completion 2027-12-20 (Estimated)

PRIMARY OUTCOMES:
to analyze the prognostic value of the phenotypes "frail and sarcopenic," "frail only," "sarcopenic only," and "robust" on the outcomes of patients with fibrosing ILDs | 12 months
  association between the classifications "non-frail," "frail" (according to the Fried score- percentage of patients), "sarcopenic" (based on EWGSOP criteria - percebntage of patients), and "frail and sarcopenic" at the initial evaluation of ILD (percentage of patients)
to analyze the progression of sarcopenia | up to 12 months
  composite outcome comprising death, hospitalization, or progression of fibrosing ILD (percentage of patients)

IPD SHARING:
Plan to Share IPD: No